CLINICAL TRIAL: NCT06761183
Title: Safety and Preliminary Efficacy of NXL-001 in Patients with Ischemic Stroke
Acronym: NXL-001
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, yilong Wang, Chief physician, Professor, Beijing Tiantan Hospital
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: KY2024-378-02
Record Dates: First submitted 2024-12-27; First posted 2025-01-07 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2024-12

CONDITIONS: Ischemic Stroke
Keywords: Ischemic Stroke; Gene therapy
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Intervention Model Description: intracerebral stereotactic injection of NXL-001：with 3 subjects in each group to receive a single stereo-tactically intracerebral injection of NXL-001 at escalating doses.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- intracerebral stereotactic injection of NXL-001 (Experimental): intracerebral stereotactic injection of NXL-001: with 3 subjects in each group to receive a single stereo-tactically intracerebral injection of NXL-001 at escalating doses.
  Interventions: Genetic: intracerebral stereotactic injection of NXL-001

INTERVENTIONS:
Genetic: intracerebral stereotactic injection of NXL-001 — intracerebral stereotactic injection of NXL-001: with 3 subjects in each group to receive a single stereo-tactically intracerebral injection of NXL-001 at escalating doses.

SUMMARY:
This is a single-arm, open-label, single center, dose-escalation exploratory clinical study to evaluate the safety and tolerability of a single intracerebral injection of NXL-001, a NeuroD1 base gene therapy, in patients with chronic neuronal deficits from ischemic stroke.

DETAILED DESCRIPTION:
The death of neurons after stroke is the direct cause of brain function loss, and the difficulty of neurons to regenerate themselves in the adult brain is an important reason for the lack of effective treatment for stroke. Replacing the lost neurons and then reconstructing the functional connectivity between neurons is the key to improving stroke symptoms. NXL-001 is a gene therapy, using an AAV9 (adeno-associated virus 9) vector to deliver and express the neurodevelopmental transcription factor NeuroD1 to directly convert astrocytes into functional neurons. NXL-001 has been shown to regenerate neurons and improve motor function when administered in animal models of stroke. The primary objective of this single-arm, open-label, single center, dose-escalation study is to evaluate the safety and tolerability of intracerebral stereotactic injection of NXL-001. The secondary objective is to preliminarily evaluate the efficacy of NXL-001 in patients with chronic neuronal deficits from ischemic stroke and to determine its safe and effective dose range. This dose escalation study involves three cohorts, with 3 subjects in each group to receive a single stereo-tactically intracerebral injection of NXL-001 at escalating doses.

ELIGIBILITY:
Inclusion Criteria:

* Age 40-75 years, inclusive, gender is not limited.
* Clinical diagnosis of ischemic stroke confirmed by neuro-imaging（CT , MRI，et al）.
* 2-4 months after the onset of ischemic stroke.
* MRI scan shows that the stroke lesion is 20-80ml in size, with cerebral motor cortex injury, and DTI shows corticospinal tract injury.
* Persisting moderate to severe motor function impairment due to stroke after standardized and guide-recommended rehabilitation therapy, characterized by baseline NIHSS score of 6-20 points, and a motor score of 3-4 on the affected upper or lower limb.
* Expected survival ≥ 12 months.
* The patient or his/her legal representative clearly understands, voluntarily participates in the study and signs the informed consent form.
* The subject is willing and able to return for follow-up visits as required by the trial protocol.
* Able to undergo rehabilitation training and treatment;
* Male and female subjects participating in the clinical study must agree to use an adequate birth control method for at least 6 months after administration

Exclusion Criteria:

* Motor deficit due to ischemic stroke of posterior circulation.
* Motor deficit due to any other causes.
* History of epilepsy.
* History of encephalitis, meningitis, multiple sclerosis or other central nervous system infections.
* History of intracranial hemorrhage and subarachnoid hemorrhage.
* History of severe head trauma within the past 5 years.
* Any contraindications to MRI scanning (such as implanted pacemaker, infusion pump etc.).
* Serum anti-AAV9 antibody titers ≥ 1:100
* History of malignant tumors within 5 years before screening (except for adequately treated cervical carcinoma in situ, papillary thyroid cancer, basal cell or squamous epithelial cell skin cancer, localized prostate cancer after radical surgery, and breast ductal carcinoma in situ).
* Active infections, including but not limited to human immunodeficiency virus (HIV), hepatitis A, B or C, syphilis, etc.
* Received any investigational drugs within 3 months (or 5 half-lives of the investigational drug, whichever is longer) of initial screening.
* Received any other cell and/or gene therapy for stroke.
* Requirement for anticoagulants.
* Intermittent use of oral anti-spasticity medications (stop/start date from 1-month prior-to and 3-month post- NXL-001 administration). Use of oral anti-spasticity medications are acceptable if they have been taken regularly for at least one month prior to NXL-001 administration).
* Pregnant or lactating female subjects.
* Insufficient reserved functions of liver, kidney and bone marrow: Neutrophil count <1,500/mm 3 ; platelets <100, 000/mm 3 ; hemoglobin <9.0 g/dL; serum creatinine >1.5 times the upper limit of normal range (ULN) ; renal function eGFR < 60mL/min/ 1.73m2 ; Bilirubin, aspartate aminotransferase (AST) and alanine aminotransferase (ALT) >2.5 times ULN; activated partial prothrombin time ( APTT ) or international normalized ratio ( INR ) >1.3 times ULN.
* Poorly controlled illness judged by the investigator at screening, including cardiovascular system (decompensated heart failure (NYHA classification III and IV), unstable angina, acute myocardial infarction), Respiratory system, digestive system, endocrine metabolic system, neuropsychiatric system, blood system and immune system diseases, etc.
* Based on medical history and investigator's judgment, the subject is at significant risk of suicide.
* In the investigator's judgment, the subject has any other factors deemed inappropriate for participation in this trial.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2025-01-31 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of NXL-001 | baseline to month 3 after dose
  Incidence of adverse events (AE) and serious adverse events (SAE) according to CTCAE 5.0

SECONDARY OUTCOMES:
Change in MRI images from baseline at month 12 | Baseline (Screening), and on day 7, month 1,3,6 and 12 after dose
  Changes in MRI images of cerebral infarction areas before and after treatment
Change in PET images from baseline at month 12 | Baseline (Screening), and at month 3 and 12 after dose
  Changes in PET images will be used to assess metabolic changes in the infarct and its surrounding area before and after treatment
Change in the National Institutes of Health Stroke Scale (NIHSS) Total Score from baseline to month 12 | Baseline (Screening), and on day1, 7, and at month 1,3,6 and 12 after dose
  The NIHSS is a standardized method used to measure the level of impairment caused by a stroke. The scale consists of 11 items that measure several aspects of brain function, including consciousness, vision, sensation, movement, speech, and language. A certain number of points are given for each impairment uncovered during a focused neurological examination. A maximal score of 42 represents the most severe and devastating stroke with 0=no stroke, 1-4=minor stroke, 5-15=moderate stroke, 15-20=moderate/severe stroke, and 21-42=severe stroke.
Change in the Modified Rankin Scale (mRS) Response from Baseline to Month 12 | Baseline (Screening), and on day1, 7, and at month 1,3,6 and 12 after dose
  The mRS is a commonly used scale for measuring the degree of disability in daily activities for patients who have suffered a stroke. The mRS is an ordinal scale from 0 (no symptoms at all) to 5 (severe disability; requiring constant nursing care and attention, bedridden, incontinent) with a sixth category of death.
Change in the Fugl-Meyer Assessment (FMA) from Baseline to Month 12 | Baseline (Screening), and at month 1,3,6 and 12 after dose
  The FMA is used as a clinical measure of body function impairment after stroke that assesses several dimensions of motor impairment, including range of motion in upper and lower limbs, reflex activity, volitional movement, and coordination.The Fugl-Meyer motor total score ranged from 0 (hemiplegia) to a maximum of 100 points (normal motor performance), and is comprised of a 33-item upper extremity subscale (UE-FMMS) and the 17-item lower extremity subscale (LE-FMMS). Items were scored on a 3-point ordinal scale: 0= cannot perform; 1= partial motion; 2= full motion Individual items are summed to determine scores for the 2 subscale scores, as well as a motor total score (total of the 2 subscales UE-FMMS and LE-FMMS). As a result, the UE-FMMS subscale score ranged from 0 to 66 and the LE-FMMS subscale score ranged from 0 to 34. A maximally affected person will have a score of 0 while a fully functional person will have the highest score (i.e., 34 for LE-FMMS, 66 for UE-FMMS, 100 for FMM)
Change in the modified Ashworth Scale from baseline to month 12 | Baseline (Screening), and at month 1,3,6 and 12 after dose
  The Modified Ashworth Scale (MAS) is the most commonly used clinical scale to measure hypertonic or spastic muscle. The scale ranges from 0 to 4, with the muscle acting across the joint rated based on what point during flexion or extension resistance or a catch is noted. A score of 0 indicates no resistance to passive movement, with a 4 indicating a rigid joint.
Change in the gait function scale from baseline to month 12 | Baseline (Screening), and at month 1,3,6 and 12 after dose
  The gait function scale consists of 4 items that measure several aspects of gait function quantitatively and semi-quantitatively, including balance, Six-meter Walk test, Tandem walking test, and Quick sit-up test.
Change in the Action Research Arm Test (ARAT) from baseline to month 12 | Baseline (Screening), and at month 1,3,6 and 12 after dose
  The Action Research Arm Test (ARAT) is a 19-item observational measure to assess upper extremity performance (coordination, dexterity and functioning) in stroke recovery, brain injury and multiple sclerosis populations. Items comprising the ARAT are categorized into four subscales (grasp, grip, pinch and gross movement) and arranged in order of decreasing difficulty, with the most difficult task examined first, followed by the least difficult task. Each item is rated 4 (0-3 points), 0 = no movement；1= movement task is partially performed；2 = movement task is completed but takes abnormally long；3 = movement is performed normally. Scores on the ARAT may range from 0-57 points, with a maximum score of 57 points indicating better performance.
Change in the EQ-5D-5L scale from baseline to month 12 | Baseline (Screening), and at month 1,3,6 and 12 after dose
  The EQ-5D, EuroQol Five Dimensions Questionnaire, is a set of standardized scales measuring health status. The EQ-5D-5L descriptive system consists of five dimensions (each describing a specific aspect of health): mobility, self-care, daily activities, pain or discomfort, anxiety or depression. Each dimension has five response levels: no problems, slight problems, moderate problems, severe problems, unable to/extreme problems. The respondent is asked to indicate his/her health state by checking the box next to the most appropriate response level for each of the five dimensions.
Change in the Electroencephalogram（EEG）from baseline to month 12 | Baseline (Screening), and at month 1,3,6 and 12 after dose
  EEG is a simple, low-cost, non-invasive tool that can provide information about the changes occurring in the cerebral cortex during the recovery process after stroke. EEG provides data on the evolution of cortical activation patterns.
Change in the Motor-evoked potential (MEP) from baseline to month 12 | Baseline (Screening), and at month 1,3,6 and 12 after dose
  Motor evoked potential (MEP) amplitude and threshold are predictors of functional outcome in the early stages after stroke, and improvement in these parameters usually accompanies motor recovery.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ma NX, Puls B, Chen G. Transcriptomic analyses of NeuroD1-mediated astrocyte-to-neuron conversion. Dev Neurobiol. 2022 Jul;82(5):375-391. doi: 10.1002/dneu.22882. Epub 2022 May 23. PMID 35606902
- [Background] Kuwabara T, Hsieh J, Muotri A, Yeo G, Warashina M, Lie DC, Moore L, Nakashima K, Asashima M, Gage FH. Wnt-mediated activation of NeuroD1 and retro-elements during adult neurogenesis. Nat Neurosci. 2009 Sep;12(9):1097-105. doi: 10.1038/nn.2360. Epub 2009 Aug 23. PMID 19701198
- [Background] Wu S, Wu B, Liu M, Chen Z, Wang W, Anderson CS, Sandercock P, Wang Y, Huang Y, Cui L, Pu C, Jia J, Zhang T, Liu X, Zhang S, Xie P, Fan D, Ji X, Wong KL, Wang L; China Stroke Study Collaboration. Stroke in China: advances and challenges in epidemiology, prevention, and management. Lancet Neurol. 2019 Apr;18(4):394-405. doi: 10.1016/S1474-4422(18)30500-3. PMID 30878104
- [Background] Zerna C, Hegedus J, Hill MD. Evolving Treatments for Acute Ischemic Stroke. Circ Res. 2016 Apr 29;118(9):1425-42. doi: 10.1161/CIRCRESAHA.116.307005. PMID 27126651
- [Background] Zhou M, Wang H, Zeng X, Yin P, Zhu J, Chen W, Li X, Wang L, Wang L, Liu Y, Liu J, Zhang M, Qi J, Yu S, Afshin A, Gakidou E, Glenn S, Krish VS, Miller-Petrie MK, Mountjoy-Venning WC, Mullany EC, Redford SB, Liu H, Naghavi M, Hay SI, Wang L, Murray CJL, Liang X. Mortality, morbidity, and risk factors in China and its provinces, 1990-2017: a systematic analysis for the Global Burden of Disease Study 2017. Lancet. 2019 Sep 28;394(10204):1145-1158. doi: 10.1016/S0140-6736(19)30427-1. Epub 2019 Jun 24. PMID 31248666